CLINICAL TRIAL: NCT00611546
Title: Study of the Oxidant-Antioxidant Effects of Parenteral Nutrition in Preterm Neonates
Brief Title: Perenteral Nutrition and Oxidative Stress in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Nehad Nasef, Mansoura University Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003-MD-thesis-nehad
Record Dates: First submitted 2008-01-24; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Preterm Infants
Keywords: preterm; parenteral nutrition; TPN; lipid emulsions; photo-protection; oxidative stress
MeSH Terms: conditions — Premature Birth; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Perenteral nutrition bottle and tubing are not protected from light
  Interventions: Other: Photo-exposure
- 2 (Active Comparator): Perenteral nutrition bottle and tubing are protected from light
  Interventions: Other: Photo-protection

INTERVENTIONS:
Other: Photo-protection — Parenteral solutions are protected from day light using aluminum covers
  Arms: 2
Other: Photo-exposure — Perenteral nutrition bottles and tubings are allowed to be exposed to day light.
  Arms: 1

SUMMARY:
In an effort to decrease the load of peroxides in TPN solutions, multiple studies examined different strategies such as photo-protection, adding multivitamins to the lipid emulsion rather than to the dextrose-amino acid admixture, and adding antioxidants such as glutathione to the TPN solution. However, the role of trace elements as antioxidants, and their interaction with light have not been studied. Also, the impact of TPN-related oxidants on clinical morbidities has not been addressed. Therefore, we aimed in this study of preterm infants to evaluate the role of different components of TPN on urinary peroxides and to examine the biochemical and clinical effects of light protection.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants included are:

1. with gestational age between 28 to 34 weeks
2. managed with TPN as part of their care in the NICU
3. their postnatal age on enrolment was < 7 days

Exclusion Criteria:

Infants are excluded if they have:

1. Clinical evidence of sepsis, or a positive blood culture on admission
2. Hepatobiliary dysfunction
3. Persistent metabolic acidosis with base deficit > 10 mEq / L
4. Renal impairment (urine output < 1 ml/kg/hour and serum creatinine > 1 mg/dl)
5. Disseminated intravascular coagulopathy
6. Maternal conditions known to be associated with oxidative stress such as preeclampsia, hypertension and diabetes.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2003-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Concentration of peroxides in the urine | 48 hours

SECONDARY OUTCOMES:
Clinical morbidities (death, and bronchopulmonary dysplasia) | during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Bassiouny, MD, Study Chair — Mansoura University Children's Hospital

REFERENCES:
- [Derived] Bassiouny MR, Almarsafawy H, Abdel-Hady H, Nasef N, Hammad TA, Aly H. A randomized controlled trial on parenteral nutrition, oxidative stress, and chronic lung diseases in preterm infants. J Pediatr Gastroenterol Nutr. 2009 Mar;48(3):363-9. doi: 10.1097/mpg.0b013e31818c8623. PMID 19274793